CLINICAL TRIAL: NCT06121284
Title: A Randomized Placebo-controlled Trial of Adjunctive D-Cycloserine and Accelerated Intermittent Theta Burst Stimulation for Emerging Adults With Suicidal Ideation
Brief Title: iTBS+D-Cycloserine for Youth Suicide
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: REB22-1115
Record Dates: First submitted 2023-08-25; First posted 2023-11-07 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Suicidal Ideation; Suicide, Attempted; Depression, Anxiety
Keywords: Transcranial Magnetic Stimulation; Emerging Adults; Youth; Suicidal Ideation; Depression; D-Cycloserine; Cognition
MeSH Terms: conditions — Suicidal Ideation; Suicide, Attempted; Depression; Anxiety Disorders | interventions — Cycloserine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- D-Cycloserine (Experimental): Participants will orally ingest a standard 100mg dose of D-Cycloserine daily (Monday-Friday) during 2 weeks of accelerated rTMS treatments (20 sessions; 2 sessions/day separated by 1 hour). D-Cycloserine will be ingested 60-120 minutes prior to the first rTMS treatment of the day.
  Interventions: Drug: D-Cycloserine; Device: intermittent Theta-Burst-repetitive Transcranial Magnetic Stimulation
- Placebo (Placebo Comparator): Participants will orally ingest a standard 100mg dose of a microcrystalline placebo capsule daily (Monday-Friday) during 2 weeks of accelerated rTMS treatments (20 sessions; 2 sessions/day separated by 1 hour). The Placebo will be ingested 60-120 minutes prior to the first rTMS treatment of the day.
  Interventions: Device: intermittent Theta-Burst-repetitive Transcranial Magnetic Stimulation; Drug: Placebo oral tablet

INTERVENTIONS:
Drug: D-Cycloserine — Participants will orally ingest a capsule containing a 100mg dose of the antibiotic d-cycloserine daily (Monday-Friday) during 2 weeks of twice daily rTMS treatment (20 sessions) 60-120 minutes prior to the first rTMS treatment of the day.
  Arms: D-Cycloserine
Device: intermittent Theta-Burst-repetitive Transcranial Magnetic Stimulation — Repetitive Transcranial magnetic stimulation (rTMS) will be delivered using a MagPro X100 device with B70 coil and the intermittent theta burst (iTBS) protocol to the left dorsolateral prefrontal cortex. Participants will receive twice daily treatments (Monday-Friday) over two weeks (20-sessions).
Drug: Placebo oral tablet — Participants will orally ingest a capsule identical to that containing the study medication, however, this capsule will contain a placebo. They will ingest this capsule daily (Monday-Friday) for 2 weeks of twice-daily rTMS treatment (20 sessions) 60 - 120 minutes prior to the first rTMS treatment of the day.
  Arms: Placebo

SUMMARY:
Background and Rationale: Suicide is the second leading cause of death in Canadian Emerging Adults (EAs; 18-24yrs). Current treatments for suicidal thoughts and behaviors are limited and novel treatments are required to save lives. Transcranial Magnetic Stimulation (TMS) is a non-invasive neurostimulation treatment for major depressive disorder, a mental health condition at high risk for suicide. It is well tolerated and effective. However, in the child and youth population, it does not appear to be superior to sham-TMS. Therefore, strategies for enhancing TMS outcomes are required.

Over time, TMS can change the function of brain regions important in depression to reduce the symptoms of depression, including suicidal ideation. The investigators believe this occurs through a process called 'synaptic plasticity', or the process by which neurons change their connectivity with other neurons in an activity-dependent manner. Using an adjunct to facilitate these changes in the EA population may improve TMS outcomes, including both implicit and explicit measures of suicide risk.

The investigators' previous data indicates that, in adults, the effects of a TMS protocol called intermittent theta-burst stimulation (iTBS) can be enhanced by pairing stimulation with a medication called D-Cycloserine. This FDA-approved medication leads to enhanced synaptic plasticity with iTBS. In adults, this combination led to greater improvements in depression symptoms and both implicit and explicit suicide risk. Implicit suicide risk is measured with a computerized test, called the death/suicide implicit association test (Death/Suicide IAT), and explicit suicide risk is defined as suicidal thoughts reported by the individual.

In the current study, we aim to determine whether the effects of iTBS can be augmented with D-Cycloserine to reduce suicide risk in the EA population. Typical courses of iTBS involve daily treatments over 6 weeks, a timeframe that is not acceptable in individuals experiencing suicidal ideation. For this reason, we will build on data indicating that treatment courses can be condensed by delivering multiple treatments in a single day to accelerate symptomatic improvements. Specifically, our data suggests that (1) 4-weeks of daily iTBS+D-Cycloserine significantly improves implicit and explicit suicide risk and (2) a single-dose of D-Cycloserine paired with two iTBS treatments separated by one hour, enhances the physiological effects of iTBS. As such, in this study, participants will receive two treatments per day, separated by an hour, thereby accelerating a typical 4-week course to 2 weeks.

Research Question and Objectives: To conduct a 2-week double-blind placebo-controlled randomized clinical trial where 54 participants will be randomly assigned to one of two groups: 1) accelerated iTBS+D-Cycloserine, and 2) accelerated iTBS+placebo. The primary outcome of the study is performance on the Death/Suicide-IAT, a measure of suicide risk; however, we will also determine whether pairing stimulation with D-Cycloserine enhances the antidepressant effects of iTBS, reduces suicidal ideation in this population, and reduces the likelihood of engaging in suicidal behavior or having suicidal crises over the following six months.

DETAILED DESCRIPTION:
Methods: 54 participants between 18-24 years old with clinically significant past week suicidal ideation, defined as a score ≥4 on item 10 of the Montgomery Asberg Depression Rating Scale (MADRS), at least moderate depressive symptoms (≥15 Hamilton Depression Rating Scale-17 [HAMD-17]), and a history of at least one suicide attempt will be recruited. It is important to note that suicidal ideation occurs on a spectrum and that scores on the MADRS item 10 range from 0-6. A score of 4 = "Probably better off dead. Suicidal thoughts are common, and suicide is considered as a possible solution, but without specific plans or intention." A score of 6 = "Explicit plans for suicide when there is an opportunity. Active preparations for suicide." Within this range, an individual may have active or passive suicidal ideation with or without intent or a plan. Individuals with active suicidal ideation, intent, or plan will be eligible to participate in the study if they are currently admitted as an inpatient.

Participants will complete a screening visit to determine eligibility based on the inclusion/exclusion criteria. If the participants are not eligible, no further study procedures will be conducted. Eligible subjects will be randomized in a 1:1 ratio to receive either accelerated iTBS+placebo or accelerated iTBS+D-Cycloserine. The randomization sequence will be generated with random number generation, a block size of 6, and allocation concealment.

Double-blind assignment and allocation concealment will be maintained by sequential numbering. Patients will be randomly assigned to receive either accelerated iTBS+D-Cycloserine or accelerated iTBS+placebo treatments. Patients without blood work within the past month will have laboratory tests done to rule out hematological, hepatic, and renal disease.

The primary outcome of interest is change in performance on the Death/Suicide-IAT from baseline to treatment end. Performance on this measure and other cognitive tasks will also be assessed at 1-month and 6-month follow-ups.

Clinical outcomes will be quantified using change on the clinician-rated Scale for Suicidal Ideation (SSI) and MADRS and self-reported measures of depression and anxiety. These symptoms will be assessed at baseline, week-1 (halfway), week-2 (end of treatment), one month, and 6-months post-treatment. Change in suicidal behaviors over the 6-months prior and following treatment will also be assessed using the Columbia Suicide Severity Rating Scale (CSSRS) and medical record review.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals aged 18 to 24 years
2. Any sex or gender
3. Are competent to consent to treatment
4. Have previously attempted suicide as defined by the Columbia Suicide Severity Rating Scale
5. Currently have suicidal ideation as defined by a score ≥4 on item 10 of the MADRS in the past week. Individuals with active suicidal ideation, defined as suicidal ideation with the intention to act on a plan that might result in death, are only eligible if currently hospitalized
6. Moderate depression measured on the 17-item Hamilton Rating Scale for Depression (HAMD-17) ≥15
7. Are able to adhere to the treatment schedule
8. Pass the TMS adult safety screening (TASS) questionnaire
9. Have a normal ECG, CBC, electrolytes, BUN, creatinine, eGFR, AST, ALT, and GGT within the last month.

Exclusion Criteria:

1. Allergy to cycloserine or any excipients due to possible anaphylaxis or other reactions.
2. Current alcohol or substance misuse.
3. Current symptoms or history of psychosis, as this can be aggravated by D-Cycloserine.
4. Are currently pregnant, breast feeding or plan to become pregnant during the study, as the effects of D-Cycloserine on the fetus are unknown. Health Canada requires that women of reproductive potential utilize either highly effective birth control or double barrier method of contraception. Abstinence is only acceptable when it is the usual and preferred lifestyle of the participant.
5. Have failed a course of ECT in the current episode. Previous ECT treatment outside of the current episode does not influence inclusion.
6. Have previously failed a course of rTMS treatment
7. Have any significant neurological disorder or insult as this increased the risk of adverse events with rTMS including, but not limited to any condition likely to be associated with increased intracranial pressure, space occupying brain lesion, any history of epilepsy, cerebral aneurysm, Parkinson's disease, Huntington's chorea, multiple sclerosis, significant head trauma with loss of consciousness for greater than or equal to 15 minutes
8. Have concomitant major unstable medical illness, cardiac pacemaker or implanted medication pump
9. Have an intracranial implant (e.g., aneurysm clips, shunts, stimulators, cochlear implants, or electrodes) or any other metal object within or near the head, excluding the mouth, that cannot be safely removed because these can heat or move due to the rapidly alternating magnetic field generated by rTMS.
10. Are currently being treated with GABA agonists such as benzodiazepines, cyclopyrrolones, gabapentin/pregabalin, or anticonvulsant due to the potential to limit TMS efficacy
11. Those with a history of intracranial implants or metal, or with any potential metal fragments in the body (particularly in the orbits).

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 54 (Estimated)
Dates: Start 2024-03-11 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Performance on the Death Implicit Association Test (D-IAT) at treatment end | Change from baseline to end of treatment (week 2)
  The D-IAT measures reaction time in categorizing life and death-related words. Different pairings of target attributes (Life/Death) and attribute dimensions (Me/Not Me) create implicit associations between the self with life and death. The D-IAT score is interpreted as a difference in strength of implicit association of the self with life and death. Scores range from -2 (strong implicit association with life) to +2 (strong implicit association with death).

SECONDARY OUTCOMES:
Performance on the Death Implicit Association Test (D-IAT) at follow up | Baseline, treatment end (2-weeks), 1-month, 6-months
  The D-IAT measures reaction time in categorizing life and death-related words. Different pairings of target attributes (Life/Death) and attribute dimensions (Me/Not Me) create implicit associations between the self with life and death. The D-IAT score is interpreted as a difference in strength of implicit association of the self with life and death. Scores range from -2 (strong implicit association with life) to +2 (strong implicit association with death).
Change on the Scale for Suicidal Ideation (SSI) at end of treatment (week 2) | SSI score from baseline to end of treatment (week 2)
  Change in score on the clinician administered SSI. This consists of 19 items rated on a Likert-scale from 0 to 2. Higher scores are indicative of worse suicidal ideation.
SSI at 1-month post treatment | SSI score at 1-month post treatment
  Score on the clinician-administered SSI. This consists of 19 items rated on a Likert scale from 0 to 2. Higher scores are indicative of worse suicidal ideation.
SSI at 6-months post treatment | Administered at 6-months post treatment
  Score on the clinician administered SSI. This consists of 19 items rated on a Likert-scale from 0 to 2. Higher scores are indicative of worse suicidal ideation.
Change on the Montgomery Asberg Depression Rating Scale (MADRS) post treatment | MADRS score at week 2 (post treatment)
  Change in severity of depressive symptoms as measured by the MADRS, a clinician-rated instrument. The MADRS is a ten-item diagnostic questionnaire used to measure the severity of depressive episodes. The overall score ranges from 0 - 60. Cutoff points are 0-6 = normal, 7-9 = mild depression, 20-34 = moderate depression, >34 = severe depression.
Montgomery Asberg Depression Rating Scale (MADRS) at 1-month | MADRS score at 1-month follow up
  Severity of depressive symptoms as measured by the MADRS, a clinician-rated instrument. The MADRS is a ten-item diagnostic questionnaire used to measure the severity of depressive episodes. The overall score ranges from 0 - 60. Cutoff points are 0-6 = normal, 7-9 = mild depression, 20-34 = moderate depression, >34 = severe depression.
Montgomery Asberg Depression Rating Scale (MADRS) at 6-months | MADRS score assessed at 6-month follow up
  Severity of depressive symptoms as measured by the MADRS, a clinician-rated instrument. The MADRS is a ten-item diagnostic questionnaire used to measure the severity of depressive episodes. The overall score ranges from 0 - 60. Cutoff points are 0-6 = normal, 7-9 = mild depression, 20-34 = moderate depression, >34 = severe depression.
Clinical Global Impression (CGI) - Severity | The CGI will be administerd at baseline, week 1, week 2 (end of treatment), 1-month follow up (week 6), and 6-month follow up.
  The CGI-Severity scale is clinician rated from 1-7 representing 'Not at all ill' to 'Severely ill'.
Clinical Global Impression (CGI) - Improvement | The CGI will be administerd at baseline, week 1, week 2 (end of treatment), 1-month follow up (week 6), and 6-month follow up.
  The CGI-Severity scale is clinician rated from 1-7 representing 'Not at all ill' to 'Severely ill'.
Change on the Borderline Symptom List-23 (BSL-23) | The BSL-23 will be completed at baseline, week 2 (end of treatment), 1-month, and 6-month follow up visits
  The BSL is a self-report measure of 23 questions assessing symptoms of borderline personality disorder on a Likert scale from 0-4.
Self-Reported Quick Inventory of Depressive Symptoms (QIDS-SR) | The QIDS-SR will be completed at baseline, week 2, 1-month, and 6-month follow up visits.
  The Quick Inventory of Depressive Symptomatology (QIDS) rates depression symptoms via self-assessment.Severity of depression can be judged based on the total score.
  1-5 = No depression 6-10 = Mild depression 11-15 = Moderate depression 16-20 = Severe depression 21-27 = Very severe depression
Generalized Anxiety Disorder-7 item questionnaire (GAD-7) | The GAD-7 will be completed at baseline, week 2, 1-month, and 6-month follow up visits.
  Anxiety symptoms will be assessed using the 7 item Generalized Anxiety Disorder (GAD-7) questionnaire. The GAD-7 measures self-reported feelings of anxiety within the last 2 weeks. Scores range from 0-21. Scores of 5, 10, and 15 represent cut points for mild, moderate, and severe anxiety, respectively.
Difficulties in Emotional Regulation Scale (DERS) | The DERS will be completed at baseline, week 2, 1-month, and 6-month follow up visits.
  The DERS is a 36-item self-reported measure of emotional regulation ability, rated on a Likert-Scale from 0 (almost never) to 5 (almost always).
WHO Quality of Life Questionnaire (WHOQOL-BREF) | The WHOQOL-BREF will be completed at baseline, week 2, 1-month, and 6-month follow up visits.
  The WHOQOL-BREF is a self-reported questionnaire which assesses individual's perception of their quality of life across 4 domains; physical health, psychological, social relationships and environment. Domains scores are calculated to range from 0-20 and scaled in a positive direction (ie. higher scores denote higher quality of life).
Beck Hopelessness Scale (BHS) | The BHS will be completed at baseline, week 2, 1-month, and 6-month follow up visits.
  The BHS is a self-reported measure of hopelessness that includes 20 true/false questions that assess three different aspects of hopelessness: feelings about the future, loss of motivation, and future expectations. Higher scores reflect higher levels of hopelessness.
Performance on the Spatial Working Memory Task (SWM; CANTAB) | the SWM task will be completed at baseline, week 2 (end of treatment), 1-month, and 6-month follow up
  The SWM task requires the retention and manipulation of visuo-spatial information. It acts as a measure of strategy and errors when using spatial working memory.
Performance on the Stroop Word-Colour Task (SWCT) | The SWCT will be completed at baseline, week 2 (end of treatment), 1-month and 6-month follow up
  The SWCT is a measure of cognitive control which uses reaction times to assess an individual's ability to inhibit a pre-potent response.
Performance on the Intra-Extra Dimensional Set Shift (IED; CANTAB) | The IED will be completed at baseline, week 2 (end of treatment), 1-month, and 6-month follow up
  The IED measures an individual's ability to understand and apply the rules of a game as the rules change (acquisition and reversal).
Suicidal behaviors over 6-months post-treatment | Columbia Suicide Severity Rating Scale and electronic medical record verification assessed 6-months post treatment
  Suicide attempts, aborted suicide attempts, interrupted suicide attempts, suicidal ideation and non-suicidal self-injury will be measured using the Columbia Suicide Severity Rating Scale (CSSRS). Higher scores on the CSSRS are indicative of more severe suicidal behaviors.
Change in psychiatric emergency department visits and hospitalizations over 6 months pre and post-treatment | The medical record will be accessed six months after the completion of treatment.
  Participants' medical record will be reviewed for emergency department presentations for a psychiatric chief complaint and psychiatric hospitalizations in the six months prior to and following treatment.

OTHER OUTCOMES:
Incidence of Treatment Emergent Adverse Events | Daily (monday-friday) throughout 2-weeks of treatment, at 1-month, and 6-months post treatment
  Adverse events will be tracked and recorded
Side Effects | The TSES will be administered at baseline, end of week 1 (halfway), and end of week 2 (end of treatment)
  Side effects will be tracked through the Toronto Side Effects Scale (TSES). The TSES is a self reported questionnaire that assesses incidence, frequency, and severity of central nervous system, gastrointestinal, and sexual side effects. Individuals will be asked to rate frequency of each symptom within the last week on a 5-point scale, from "Never" (1) to "Everyday" (5). Severity of each symptom is similarly rated on a 5-point scale, from "No trouble" (1) to "Extreme Trouble" (5).
Complete Blood Count (CBC): Hemoglobin | Screening and end of treatment (end of week 2)
  A complete blood count (CBC) panel will be used to measure the amount of hemoglobin present in the blood from a whole blood sample, measured in g/L. Results must be within the normal reference range prior to entering the study. Results from the baseline and treatment end will be compared with paired t-tests.
Complete Blood Count (CBC): Hematocrit | Screening and end of treatment (end of week 2)
  A complete blood count (CBC) panel will be used to measure the amount of hematocrit present in the blood from a whole blood sample, measured in L/L. Results must be within the normal reference range prior to entering the study. Results from the baseline and treatment end will be compared with paired t-tests.
Complete Blood Count (CBC): White Blood Cell Count (WBC) | Screening and end of treatment (end of week 2)
  A complete blood count (CBC) panel will be used to measure the amount of white blood cells (WBC) present in the blood from a whole blood sample, measured in 10^9/L. Results must be within the normal reference range prior to entering the study. Results from the baseline and treatment end will be compared with paired t-tests.
Complete Blood Count (CBC): Red Blood Cell count (RBC) | Screening and end of treatment (end of week 2)
  A complete blood count (CBC) panel will be used to measure the amount of red blood cells (RBC) present in the blood from a whole blood sample, measured in 10^12/L. Results must be within the normal reference range prior to entering the study. Results from the baseline and treatment end will be compared with paired t-tests.
Complete Blood Count (CBC): Platelets | Screening and end of treatment (end of week 2)
  A complete blood count (CBC) panel will be used to measure the amount of platelets present in the blood from a whole blood sample, measured in 10^9/L. Results must be within the normal reference range prior to entering the study. Results from the baseline and treatment end will be compared with paired t-tests.
Electrolyte Panel: Sodium Level | Screening and end of treatment (end of week 2)
  An electrolyte panel will be used to measure the amount of sodium present in the blood from a whole blood sample, measured in mmol/L. Results must be within normal reference range prior to entering the study. Results from baseline and treatment end (end of week 2) will be compared with paired t-tests.
Electrolyte Panel: Potassium Level | Screening and end of treatment (end of week 2)
  An electrolyte panel will be used to measure the amount of potassium present in the blood from a whole blood sample, measured in mmol/L. Results must be within the normal reference range prior to entering the study. Results from the baseline and treatment end will be compared with paired t-tests.
Electrolyte Panel: Chloride Level | Screening and end of treatment (end of week 2)
  An electrolyte panel will be used to measure the amount of chloride present in the blood from a whole blood sample, measured in mmol/L. Results must be within the normal reference range prior to entering the study. Results from the baseline and treatment end will be compared with paired t-tests.
Bloodwork: Blood Urea Nitrogen (BUN) Test | Screening and end of treatment (end of week 2)
  A BUN test (aka blood urea nitrogen test) measures the level of urea nitrogen present in the blood from a whole blood sample, measured in mmol/L. Results must be within normal reference range prior to entering the study. Results from baseline and treatment end will be compared with paired t-tests.
Bloodwork: Creatinine | Screening and end of treatment (end of week 2)
  A creatinine blood test measures the level of creatinine present in the blood from a whole blood sample, measured in umol/L. Results must be within the normal reference range prior to entering the study. Results from the baseline and treatment end will be compared with paired t-tests.
Bloodwork: estimated Glomerular Filtration Rate (eGFR) Test | Screening and end of treatment (end of week 2)
  In adults, glomerular filtration rate can be easily estimated using the CKD-EPI GFR equation.
  This formula uses the patient's age and gender with the measured blood creatinine value to estimate glomerular filtration rate, or eGFR. eGFR is measured in mL/min/1.73m^2.
  Results must be within normal reference range prior to entering the study. Results from baseline and treatment end will be compared with paired t-tests.
Bloodwork: Gamma Glutamyl Transferase Test | Screening and end of treatment (end of week 2)
  A GGT test measures the level of gamma-glutamyl transpeptidase (GGT) present in the blood from a whole blood sample, measured in U/L. Results must be within the normal reference range prior to entering the study. Results from the baseline and treatment end will be compared with paired t-tests.
Bloodwork: Alanine Transaminase (ALT) | Screening and end of treatment (end of week 2)
  An ALT test measures the level of alanine transaminase (ALT) present in the blood from a whole blood sample, measured in U/L. Results must be within normal reference range prior to entering the study. Results from baseline and treatment end will be compared with paired t-tests.
Bloodwork: Aspartate Aminotransferase (AST) | Screening and end of treatment (end of week 2)
  An AST test measures the level of aspartate aminotransferase (AST) present in the blood from a whole blood sample, measured in U/L. Results must be within the normal reference range prior to entering the study. Results from the baseline and treatment end will be compared with paired t-tests.
Electrocardiogram (ECG): Heart Rate | Screening visit and end of treatment (end of week 2)
  An ECG will be completed at baseline and post-treatment (Week 2). ECG measurements will include heart rate. Results must be within the normal range prior to entering the study. Heart rate will be compared at baseline and end of treatment using paired t-tests.
Electrocardiogram (ECG): PR Interval | Screening visit and end of treatment (end of week 2)
  An ECG will be completed at baseline and post-treatment (Week 2). ECG measurements will include the PR interval is calculated from the onset of the P wave to the start of the QRS complex and reflect conduction through the AV node. Results must be within the normal range prior to entering the study. the PR interval from baseline to treatment end will be compared with paired t-tests.
Electrocardiogram (ECG): QRS Interval | Screening visit and end of treatment (end of week 2)
  An ECG will be completed at baseline and post-treatment (Week 2). ECG measurements will include QRS interval (duration) is a measurement of the time it takes for electrical activity to travel through the ventricular myocardium. The QRS interval must be within the normal range prior to entering the study. The duration of the QRS interval at baseline and end of treatment will be compared with paired t-tests.
Electrocardiogram (ECG): QTc Interval | Screening visit and end of treatment (end of week 2)
  An ECG will be completed at baseline and post-treatment (Week 2). The QT interval is calculated as the time from the start of the Q wave to the end of the T wave. The QT interval is corrected for heart rate (QTc), a process performed automatically by modern ECG recorders. Results must be within the normal range prior to entering the study. QTc from baseline to treatment end will be compared with paired t-tests.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander McGirr, MD PhD, Principal Investigator — University of Calgary
Locations (1):
- University of Calgary, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No